CLINICAL TRIAL: NCT02612103
Title: Evaluation of Markers of the Extracellular Matrix Turnover as Biomarkers in Inflammatory Bowel Diseases and Establishment of an Inflammatory Bowel Diseases (IBD) Biobank
Brief Title: Biomarkers in Inflammatory Bowel Diseases
Status: Completed | Type: Observational
Sponsor: Line Elberg Godskesen (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Line Elberg Godskesen, MD, PhD-student, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: S-20150107
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2018-03

CONDITIONS: Inflammatory Bowel Disease; Colitis, Ulcerative; Crohn Disease
Keywords: Biochemical markers
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Active Crohns disease: Verified Crohns disease diagnosis according to clinical, endoscopic and histological standard criteria and Harvey Bradshaw index > 4.
- Crohns disease in remission: Verified Crohns disease diagnosis according to clinical, endoscopic and histological standard criteria and Harvey Bradshaw index ≤ 4.
- Active ulcerative colitis: Verified ulcerative colitis diagnosis according to clinical, endoscopic and histological standard criteria and Simple Clinical Colitis Activity Index > 3.
- Ulcerative colitis in remission: Verified ulcerative colitis diagnosis according to clinical, endoscopic and histological standard criteria and Simple Clinical Colitis Activity Index ≤ 3.
- Irritable bowel syndrome: Verified irritable bowel syndrome according to standard criteria.
- Healthy controls: No known chronic diseases which needs continuously medication.

SUMMARY:
Ulcerative colitis (UC) and Crohn's disease (CD) are chronic relapsing inflammatory bowel diseases (IBD). At the time of diagnosis it is not possible to predict the course of the disease, which can range from a few flares in a lifetime to uncontrollable disease leading to hospitalization, surgery and stoma. There is a continuous need to improve diagnostic and prognostic tools.

In chronic inflammation diseases there is an excessive turnover of the extracellular tissue. Tissue is broken down to small fragments and released into the circulation. Changes in the amount of these fragments in the blood may provide information on the damage and quality of the affected tissue and may therefore act as objective measure of disease burden and severity - a so called biomarker.

The potential of such biomarkers is evaluated in a combined cross-sectional and longitudinal survey including 300 patients with UC, CD, irritable bowel disease and healthy controls. The patients are followed for up to 1 year. Changes in biomarker are correlated to standard markers of inflammation during active disease and remission.

Perspective The use of new biomarkers may offer a tool to evaluate early changes in the gut of patients with IBD, may be a supplement to the diagnosis, serve as markers for effect of treatment and prognosis, and in time be a good alternative to fecal samples or endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Written informed consent
* and one of:
* for Crohn's disease - active disease: Verified CD diagnosis according to clinical, endoscopic and histological standard criteria and Harvey Bradshaw index > 4.
* for Crohn's disease - disease in remission: Verified CD diagnosis according to clinical, endoscopic and histological standard criteria and Harvey Bradshaw index ≤ 4.
* Ulcerative colitis - active disease: Verified UC diagnosis according to clinical, endoscopic and histological standard criteria and SCCAI > 3.
* Ulcerative colitis - in remission: Verified UC diagnosis according to clinical, endoscopic and histological standard criteria and SCCAI ≤ 3.
* Irritable bowel syndrome: Verified IBS according to standard criteria.
* Healthy control: No known chronic diseases which needs continuously medication.

Exclusion Criteria:

* Common to all participants:

  * Patient with ostomy or pouch.
  * The patient has had colon cancer, dysplasia or adenomatous polyps in the colon during the recent 5 year
  * The patient is in a poor general condition.
  * The patient is pregnant at the time of inclusion or has planned pregnancy during the period of study.
  * The patient cannot understand the information material.
* Healthy control:

  * The patient has a chronic disease.
  * IBS symptoms according to standard criteria.
  * The patient has had any type of illness within the last 14 days (for example diarrhea, a cold etc.).
  * The patient has any type of on-going medication or new medication within the last 14 days (except contraceptive pills and vitamins).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: IBD and IBS patients at The Department of Medical Gastroenterology, Odense University Hospital will be asked to participate when they contact the department due to progression in disease activity or at their regular consultations in the out-patient clinic.
  Healthy controls will be recruited by advertising in local news paper and advertising in public places.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2015-11; Primary Completion 2018-01 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Serum markers of extracellular matrix proteins (C1M, C3M, C4M, C5M, P1NP, VICM, P1NP, EL-NE, BGM and Pro-C5) | Follow-up of 1 year for patients with active IBD. For all other groups the study are cross-sectional
  The biomarkers are evaluated in relation to type of disease and disease activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark